CLINICAL TRIAL: NCT05607563
Title: A Phase I Study to Evaluate the Tolerability, Safety, Pharmacokinetic Characteristics and Preliminary Efficacy of PM1009 (Anti-TIGIT/PVRIG) in Patients With Advanced Tumors
Brief Title: A Study of PM1009 (Anti-TIGIT/PVRIG) in Patients With Advanced Tumours
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Biotheus Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PM1009-A001M-ST-R
Record Dates: First submitted 2022-10-19; First posted 2022-11-07 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-11

CONDITIONS: Advanced Tumor
Keywords: PM1009; TIGIT; PVRIG

STUDY DESIGN:
Intervention Model Description: Patients sequentially receive PM1009 120 mg, 300 mg, 600 mg, 1200 mg, intravenously, Q2W
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- PM1009 120 mg monotherapy (Experimental): PM1009 120 mg
  Interventions: Drug: PM1009 injection
- PM1009 300 mg monotherapy (Experimental): PM1009 300 mg
  Interventions: Drug: PM1009 injection
- PM1009 600 mg monotherapy (Experimental): PM1009 600 mg
  Interventions: Drug: PM1009 injection
- PM1009 1200 mg monotherapy (Experimental): PM1009 1200 mg
  Interventions: Drug: PM1009 injection

INTERVENTIONS:
Drug: PM1009 injection — Participants receive PM1009 intravenously, every 2 weeks
  Other Names: PM1009

SUMMARY:
The study is being conducted to evaluate safety, tolerability, pharmacokinetics and preliminary efficacy of PM1009 for patients with advanced tumors, also to explore the recommended Phase Ⅱ Dose（RP2D） of PM1009.

PM1009 is a new novel fully human anti-TIGIT x PVRIG bispecific antibody, containing a wildtype IgG1 Fc and has high monovalent affinity to each target, it can binds to both TIGIT and PVRIG overexpressing target cells and binds to TIGIT and PVRIG simultaneously.

DETAILED DESCRIPTION:
This is a single-arm, open-label, Phase I study contains dose escalation stage and dose expansion stage.

The dose escalation stage will be following the accelerated titration design and the classic 3+3 design, with a planned enrollment of 10 to 24 patients with advanced tumors.

The dose expansion stage will be used safe and tolerable doses, with a planned enrollment of 30 patients with advanced tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients participate in the study voluntarily and sign informed consent；
* Male or female, aged 18 to 75 years (including boundary value);
* Subjects with advanced tumor confirmed by histology or cytology fail to receive standard treatment, or there is no standard treatment scheme, or standard treatment is not applicable at this stage;
* Having adequate organ function；
* ECOG score is 0-1；
* Expected survival ≥ 12 weeks；
* There is at least one assessable tumor focus.

Exclusion Criteria:

* History of severe allergic;
* Those who have received anti-TIGIT or anti-PVRIG therapy in the past;
* Patients who have grade ≥3 immune-mediated adverse event that associated with a prior immunotherapy;
* Adverse reactions to previous antitumor therapy have not recovered to NCI-CTCAE V5.0 rating ≤ 1;
* Current definite interstitial lung disease or non-infectious pneumonitis, except for local radiotherapy;
* Patients ever received the following treatments or drugs prior to the study treatment:

  1. Major organ surgery within 28 days prior to initiation of trial treatment;
  2. Received live attenuated vaccine within 28 days prior to the study treatment;
  3. Received antitumor therapy within 4 weeks prior to the study treatment;
  4. Received systemic glucocorticoid within 14 days prior to the study treatment;
* Active infection was present within 14 days before starting study treatment;
* Those with known uncontrolled parenchymal or leptomeningeal metastases;
* Patients with active autoimmune disease or a history of autoimmune disease with potential for relapse;
* Patients with other active malignancies within 5 years prior to initiation of study treatment, except for locally treatable and cured malignancies;
* History of severe cardiovascular and cerebrovascular diseases;
* Patients with uncontrolled tumor-related pain;
* Current presence of uncontrolled pleural, pericardial, and peritoneal effusions;
* History of allogeneic hematopoietic stem cell transplantation or allogeneic organ transplantation;
* History of alcohol, psychotropic substance or drug abuse;
* History of psychiatric disorders or poor compliance;
* History of immunodeficiency, including a positive HIV antibody test;
* Patients with active syphilis infection;
* Patients with active hepatitis B or C;
* Pregnant or lactating women;
* Other conditions considered unsuitable for this study by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2022-11-21 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Dose Limited Toxicity（DLT） | up to 21 days
  Occurrence of DLT after receiving PM1009 injection

SECONDARY OUTCOMES:
Recommended Phase II Dose (RP2D) | Up to 30 days after last treatment
  To determine the RP2D of PM1009 injection
Maximum observed concentration (Cmax) | Up to 30 days after last treatment
  To evaluate the Cmax of PM1009 monotherapy
Time to Cmax (Tmax) | Up to 30 days after last treatment
  To evaluate the Tmax of PM1009 monotherapy
Minimum observed concentration (Cmin) | Up to 30 days after last treatment
  To evaluate the Cmin of PM1009 monotherapy
Trough concentrations (Ctrough) | Up to 30 days after last treatment
  To evaluate the Ctrough of PM1009 monotherapy
Area under the concentration-time curve (AUC0-last) | Up to 30 days after last treatment
  To evaluate the AUC0-last of PM1009 monotherapy
AUC to the end of the dosing period(AUC0-tau) | Up to 30 days after last treatment
  To evaluate the AUC0-tau of PM1009 monotherapy
Apparent terminal elimination half-life (t1/2) | Up to 30 days after last treatment
  To evaluate the t1/2 of PM1009 monotherapy
Accumulation ratio calculated based on Cmax (Rac_Cmax) | Up to 30 days after last treatment
  To evaluate the Rac_Cmax of PM1009 monotherapy
Accumulation ratio calculated based on AUC (Rac_AUC) | Up to 30 days after last treatment
  To evaluate the Rac_AUC of PM1009 monotherapy
Objective response rate (ORR) | Up to 24 months
  Defined as the number of patients with best overall response of confirmed CR or PR per RECIST 1.1 divided by the patients with at least one tumour imaging evaluation
Disease control rate (DCR) | Up to 24 months
  Defined as the percentage of patients who have achieved CR, PR, Non-CR/Non-PD, or SD in the study.
Progression-free survival (PFS) | Up to 24 months
  Defined as the time from the date of first dose of study drug to the first observation of documented disease progression per RECIST 1.1 as determined by the Investigators or death due to any cause, whichever occurs first.
Overall survival (OS) | Up to 24 months
  Defined as the time from the date of first dose of study drug to the date of documented death due to any cause.
Anti-drug antibody (ADA) | Up to 30 days after last treatment
  To evaluate the incidence of ADA to PM1009 injection
Adverse Events（AE）and Serious Adverse Events（SAE） | Up to 30 days after last treatment
  The incidence and severity of treatment-emergent adverse events (TEAEs) and treatment related adverse events (TRAEs) graded according to NCI-CTCAE v5.0

OTHER OUTCOMES:
T-lymphocyte phenotypes | Up to six cycles (each cycle is 2 weeks)
  T-lymphocyte phenotypes in peripheral blood

CONTACTS AND LOCATIONS:
Overall Officials: Ye Guo, Principal Investigator — Shanghai Orient Hospital
Locations (1):
- Shanghai Orient Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
The data will be published or presented for publications (poster, abstract, articles or papers) or maked any presentations.
Time Frame: after the trial completed
Access Criteria: NCI is committed to sharing data in accordance with NIH policy.